CLINICAL TRIAL: NCT03826602
Title: A Phase 1, Open-Label, Fixed-Sequence, Drug-Drug Interaction Study to Evaluate the Effects of Tucatinib of the Pharmacokinetics of Metformin in Healthy Male and Female Subjects
Brief Title: A Drug-Drug Interaction Study in Healthy Volunteers of the Effects of Tucatinib on Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGNTUC-020
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Drug-drug Interaction
MeSH Terms: interventions — tucatinib; Metformin; Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tucatinib plus metformin (Experimental): Tucatinib administered twice daily on Days 2-8. Metformin administered as a single dose on Days 1 and 8. Iohexol administered via IV push on Days 1 and 8
  Interventions: Drug: Tucatinib; Drug: Metformin; Drug: Iohexol

INTERVENTIONS:
Drug: Tucatinib — 150mg administered orally twice daily
Drug: Metformin — 850mg administered orally
Drug: Iohexol — 1500 mg administered intravenously (IV)

SUMMARY:
This study is being done to look at how tucatinib might affect the way another drug (metformin) works. It will look at healthy volunteers and how tucatinib affects how the body absorbs metformin. This will help us find out whether tucatinib is safe to give together with metformin. The study will also look at how tucatinib affects how the kidneys work.

DETAILED DESCRIPTION:
This is a single center, fixed-sequence, drug-drug interaction study to assess the effects of multiple oral doses of tucatinib on the pharmacokinetics of a single oral dose of metformin in healthy subjects. The primary objective of the study is to assess the effects of tucatinib on the single-dose PK of metformin. Secondary objectives of the study are to (1) assess the safety and tolerability of metformin when coadministered with tucatinib and (2) assess the effects of tucatinib on renal function using iohexol as glomerular filtration rate (GFR) marker.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status, as defined by the absence of evidence of any clinically significant findings
* Males must agree to use a barrier method of birth control and not donate sperm during study plus 30 days after last dose of study drug
* Weight of ≥60kg
* Body mass index between 18.0 and 32.0 kg/m² (inclusive)
* Ability to abstain from alcohol-, caffeine-, and xanthine-containing food and beverages from 48 hours prior to admission through study discharge
* All nonregular medication (including over-the-counter medication, health supplements, and herbal remedies) must be stopped at least 28 days prior to admission

Exclusion Criteria:

* Females who are of childbearing potential or lactating
* Males with female partners who are pregnant, lactating, or planning to become pregnant within 30 days of the study
* Use of any investigational drug or device within 30 days of study start
* Use of tobacco products within 21 days prior to admission
* Routine or chronic use of more than 3 grams of acetaminophen daily
* Strenuous activity, sunbathing, and contact sports within 72 hours prior to first admission and for the duration of the study
* Blood transfusion within 90 days of study drug administration
* History of alcoholism or drug abuse within 2 years
* History of alcohol consumption exceeding 7 drinks/week for female participants or 14 drinks/week for male subjects
* History of donation of more than 450 mL of blood within 60 days prior to dosing, or planned donation before 30 days have elapsed since intake of study drug
* Plasma or platelet donation within 7 days of initial study drug administration
* Positive screening test for Hepatitis B, Hepatitis C, or HIV 1 or 2 (human immunodeficiency virus)
* Acute or chronic metabolic acidosis, including diabetic ketoacidosis
* Renal disease or dysfunction as suggested by serum creatinine levels or abnormal creatinine clearance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of metformin | Up to 9 days
Time to maximum observed plasma concentration (tmax) of metformin | Up to 9 days
Half-life (t1/2) of metformin | Up to 9 days
Area under the plasma concentration-time curve from time 0 to the last available measurement (AUC0-last) of metformin | Up to 9 days
Area under the plasma concentration time curve to time 0 extrapolated to infinity (AUC0-inf) of metformin | Up to 9 days
Apparent volume of distribution (V2/F) of metformin | Up to 9 days
Oral clearance (CL/F) of metformin | Up to 9 days

SECONDARY OUTCOMES:
Incidence of adverse events (as assessed by AE assessments, clinical laboratory tests, physical examinations, vital signs measurements, and 12-lead electrocardiogram) | Up to 16 days
Glomerular Filtration Rate (GFR) as measured by iohexol plasma clearance | Up to 8 days

CONTACTS AND LOCATIONS:
Overall Officials: JoAl Mayor, PharmD, BCOP, Study Director — Seagen Inc.
Locations (1):
- Pharmaceutical Research Associates, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Zhang D, Taylor A, Zhao JJ, Endres CJ, Topletz-Erickson A. Population Pharmacokinetic Analysis of Tucatinib in Healthy Participants and Patients with Breast Cancer or Colorectal Cancer. Clin Pharmacokinet. 2024 Oct;63(10):1477-1487. doi: 10.1007/s40262-024-01412-0. Epub 2024 Oct 5. PMID 39368039